CLINICAL TRIAL: NCT00003103
Title: A Phase I/IIA Dose-Escalating Trial of BCL-2 Antisense (G3139) Treatment for Patients With Androgen-Independent Prostate Cancer or Other Advanced Solid Tumor Malignancies
Brief Title: Chemotherapy in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 97-096; CDR0000065836 (Registry Identifier: PDQ (Physician Data Query)); GENTA-G3139-97/01; NCI-G97-1337
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Esophageal Cancer; Head and Neck Cancer; Kidney Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; recurrent Wilms tumor and other childhood kidney tumors; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; clear cell sarcoma of the kidney; rhabdoid tumor of the kidney
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Wilms Tumor; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — oblimersen; Docetaxel

INTERVENTIONS:
Biological: oblimersen sodium
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of oblimersen in treating patients who have solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety and plasma concentration profiles of oblimersen (G3139) administered alone or in combination with docetaxel in patients with advanced solid tumors expressing the bcl-2 oncogene. II. Determine the plasma concentration profiles, maximum tolerated dose (MTD), and/or optimal biologic dose (OBD) of this treatment regimen in these patients. III. Determine the antitumor effects of G3139, at the MTD or OBD, in combination with docetaxel in patients with androgen-independent, refractory, or recurrent prostate cancer.

OUTLINE: This is a dose-escalation study of oblimersen (G3139). Phase I: Patients receive G3139 IV on days 1-5 and docetaxel IV on day 5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of G3139 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Phase II: Patients receive G3139 continuously over 21 days at one dose level below the MTD in combination with weekly docetaxel. Patients receive up to 2 more courses of therapy in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A maximum of 57 patients (42 for phase I and 15 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Phase I: Histologically proven advanced, primary, or malignant solid tumors that are refractory to standard therapy or for which no curative therapy exists Androgen-independent prostate cancer Head and neck cancers Breast cancer Non-small cell lung cancer Colorectal cancer Ovarian cancer Esophageal cancer Bladder cancer Kidney cancer Other solid tumors Metastatic disease should not require palliative treatment within 4 weeks of enrollment Phase II: Histologically proven androgen-independent prostate cancer Serum testosterone less than 30 ng/mL Failed at least one prior chemotherapy regimen Progressive Minimum of 3 rising PSA values from baseline obtained at least 1 week apart OR Two rising PSA values more than one month apart AND At least 25% increase over range of values AND PSA at least 4 ng/mL No active CNS or epidural tumor Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Not specified Menopausal status: Not specified Performance status: Karnofsky 60-100% Life expectancy: At least 6 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL SGOT less than 3 times the upper limit of normal Prothrombin time less than 14 seconds Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No New York Heart Association class III or IV cardiac disease Pulmonary: No severe debilitating pulmonary disease Other: Not pregnant or nursing Fertile patients must use effective contraception No active infection No other severe medical problems

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: Concurrent medical therapy (i.e., gonadotropin releasing hormone analogs or diethylstilbestrol) to maintain castrate levels of serum testosterone allowed No other concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Concurrent radiotherapy to localized sites of disease not being evaluated in study allowed Surgery: Not specified Other: At least 4 weeks since prior investigational anticancer therapy and recovered No concurrent intravenous antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 1997-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States